CLINICAL TRIAL: NCT00004332
Title: Study of the Effect of Growth Hormone-Releasing Hormone Antagonist on Growth Hormone Release in Acromegaly
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11890; UMMC-1016
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Acromegaly
Keywords: acromegaly; endocrine disorders; rare disease
MeSH Terms: conditions — Acromegaly; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine whether release of endogenous growth hormone (GH)-releasing hormone is involved in GH responses to clonidine, pyridostigmine, levodopa, arginine, GH-releasing peptide, insulin-induced hypoglycemia, and exercise in patients with acromegaly.

II. Determine whether endogenous GH-releasing hormone influences the maintenance of GH hypersecretion.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Growth hormone-releasing hormone antagonist (GHRH-A) is administered to volunteers and followed with 1 of these challenges: insulin, clonidine, pyridostigmine, arginine, levodopa, growth hormone-releasing peptide, or exercise. Tests are repeated with normal saline as the control; the order of administration (control vs. pharmacologic stimulation) is randomly assigned.

Patients receive GHRH-A (dose determined in volunteer study), thyrotropin-releasing hormone, and growth-releasing hormone.

All stimulation tests follow an overnight fast.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Active acromegaly with growth hormone (GH) hypersecretion confirmed within 1 month prior to entry, i.e.: Somatomedin C elevated GH not below 2 ng/mL on standard 100 g oral glucose tolerance test Postmenopausal and hypogonadal women eligible Volunteers aged 18 to 30 recruited for up to 3 stimulation tests Weight within 15% of ideal Physical exam normal No history of disease No requirement for medication No medical or mental contraindication to protocol participation, including heavy alcohol or tobacco use No pregnant women --Prior/Concurrent Therapy-- Not specified --Patient Characteristics-- Age: 18 to 65 Hematopoietic: No anemia Hepatic: No hepatic disease Renal: No renal disease Cardiovascular: No uncontrolled hypertension No heart disease Other: No requirement for replacement gonadal steroids, glucocorticoids, or thyroxine No mental illness No heavy alcohol use No tobacco use No drug abuse No medical contraindication to protocol therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148
Dates: Start 1993-05

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Barban, Study Chair — University of Michigan